CLINICAL TRIAL: NCT05447468
Title: Influence of Proximal Motor Control in Treating Lateral Epicondylitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shereen Mohamed, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/003304
Record Dates: First submitted 2022-07-01; First posted 2022-07-07 (Actual); Last update posted 2022-07-07 (Actual); Status verified 2022-07

CONDITIONS: Lateral Epicondylitis
MeSH Terms: conditions — Tennis Elbow | interventions — Ultrasonic Waves

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- scapular muscles strengthning group (Experimental): Patients in this group A will receive scapular muscles (lower trapezius, middle trapezius and serratus anterior) strengthening along with conventional physiotherapy (pulsed ultrasound, static stretching of ECRB muscle and eccentric exercises of wrist extensors) for 6 weeks.
  Interventions: Other: Strength of lower trapezius; Other: Strength of middle trapezius; Other: Strength of serratus anterior; Other: Pulsed ultrasound; Other: Stretching of extensor carpi radialis brevis muscle; Other: Eccentric exercises of wrist extensors
- conventional physiotherapy group (Active Comparator): Patients in this group B will receive conventional physiotherapy only (pulsed ultrasound, static stretching of ECRB muscle and eccentric exercises of wrist extensors) 3 sessions per week for 6 weeks.
  Interventions: Other: Pulsed ultrasound; Other: Stretching of extensor carpi radialis brevis muscle; Other: Eccentric exercises of wrist extensors

INTERVENTIONS:
Other: Strength of lower trapezius — Ask the patient to raise arm above the head with upper extremity in line with lower trapezius muscle fibers in prone position with the shoulder joint at 135 degrees. The patient will be asked to hold position 6 seconds and perform 3 sets of 10 repetitions and 3times per week for 6 weeks.
  Arms: scapular muscles strengthning group
Other: Strength of middle trapezius — Shoulder external rotation with the shoulder abducted 90ₒ and elbow flexed 90ₒ in prone position with elbow supported on the table. The patient will be asked to hold position 6 seconds and perform 3 sets of 10 repetitions and 3times per week for 6 weeks.
  Arms: scapular muscles strengthning group
Other: Strength of serratus anterior — Ask the patient to raise the arm on a wall in the plane of the scapula in standing position.
  The patient will be asked to hold position 6 seconds and perform 3 sets of 10 repetitions and 3times per week for 6 weeks.
  Arms: scapular muscles strengthning group
Other: Pulsed ultrasound — With a 20% duty cycle, frequency of 1 MHz and intensity of 1.5 w/cm² for 5 minutes 3 times per week for 6 weeks.
Other: Stretching of extensor carpi radialis brevis muscle — Put the elbow in extension, forearm in pronation and wrist in flexion with ulnar deviation. Hold for 30s and repeat 3 times with 30s rest in between. Three times per week for 6 weeks.
Other: Eccentric exercises of wrist extensors — Ask the patient to extend elbow, pronate forearm, extend wrist and then flex the wrist slowly until full flexion is achieved. Patients should apply 3 sets of 10 repetitions 3 times per week for 6 weeks.

SUMMARY:
This study will be conducted to investigate the effect of scapular muscles (lower trapezius, middle trapezius and serratus anterior) strengthening on pain, pain free hand grip strength and functional outcome added to conventional physical therapy in patients with chronic Lateral Epicondylitis.

DETAILED DESCRIPTION:
This study will try to investigate if scapular muscles strengthening have an effective role on pain, pain free hand grip strength and function when added to conventional physical therapy in patients with LE.

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms of lateral epicondylitis from at least the past 3 months.
2. Pain in at least two of the following four tests; Tomsen test, Maudsley test, Mill's test and handgrip dynamometer test.
3. Their ages range from 30-50 years old.

Exclusion Criteria:

Subjects will be excluded from the study if they have:

1. Peripheral neuropathy.
2. Lesions of upper limb nerves.
3. History of surgery in the affected elbow 6 months ago.
4. Cervical radiculopathy.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2022-07-15 (Estimated); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of change in pain intensity | at baseline and after 6 weeks of intervention
  Using Visual analouge scale (VAS), a continuous 10 cm line ranges from no pain to very severe pain which is valid and reliable tool. The patient marks on the line the point that they feel represents their pain intensity.
Assessment of change in hand grip strength | at baseline and after 6 weeks of intervention
  Patient stands with the elbow in complete extension and the shoulder and radioulnar joints in neutral rotation. Ask the patient to slowly squeeze the dynamometer and to stop the instant discomfort is first felt. It will be performed three repetitions separated by a 20-second rest interval. Average of three trials will be recorded. The measurement is valid and reliable.
Assessment of change in function | at baseline and after 6 weeks of intervention
  Using PRTEEQ. It is a 15-item self-reported questionnaire to measure perceived pain and disability in people with LE. It has three subscales: pain, usual activities and specific activities. Each of the items of the Patient rated tennis elbow evaluation questionnaire (PRTEEQ) is scored on a 0-10 scale, where 0 is 'no pain' or 'no difficulty' and10 is 'worst ever' or 'unable to do. Ask the patients to rate the pain and difficulty that they have experienced in the last week by marking the suitable response that reflects their current state. The total score ranges from 0 to 100, where high scores indicate greater pain and disability.

CONTACTS AND LOCATIONS:
Overall Officials: Shereen Mohamed, physiotherapist, Principal Investigator — shereenm34@gmail.com
Locations (1):
- Outpatient clinic, Faculty of Physical Therapy, Cairo university, Dokki, Egypt

IPD SHARING:
Plan to Share IPD: Undecided